CLINICAL TRIAL: NCT01007084
Title: Phase IIB Study: TRAUMA HELP: Healing and Analgesia With Propranolol
Brief Title: TRAUMA HELP: Healing and Analgesia With Propranolol
Acronym: TRAUMA_HELP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of eligible patient recruits/feasibility considerations.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Samuel McLean, MD, Principle Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-1391
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Trauma
Keywords: pain; trauma; propranolol
MeSH Terms: conditions — Wounds and Injuries; Pain | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental)
  Interventions: Drug: Propranolol; Drug: Propranolol ER
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pills

INTERVENTIONS:
Drug: Propranolol — 40 mg
  Other Names: Inderal; Innopran
  Arms: Propranolol
Drug: Propranolol ER — 120 mg twice per day
  Other Names: Inderal; Innopran
  Arms: Propranolol
Drug: Sugar pills — sugar pill
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether propranolol can decrease pain symptoms in a common subset of patients admitted to a trauma center after injury.

DETAILED DESCRIPTION:
The main purpose of this pilot study is to investigate Propranolol's utility in the trauma population. Specifically, to see if it reduces pain scores post-injury.

ELIGIBILITY:
Inclusion Criteria:

* at least one fracture
* ages 18-60 yrs
* pain score >= 4
* speak and read English

Exclusion Criteria:

* gunshot, stab wound, or assault
* paraplegia/quadriplegia
* pregnancy
* psychotic, suicidal, or homicidal
* hepatic, kidney failure
* clinically unstable or intubated at time of recruitment
* hyperthyroidism
* propranolol use within the last 6 months
* significant bradycardia
* cancer (except basal cell)
* peripheral vascular disease
* heart block > 1 degree
* breastfeeding
* congestive heart failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Daily average pain score (0-10 numeric rating pain score recorded daily from patient) after study drug initiation. | Study days 1, 3, 5, 7, 10, 13, 17, and 19

SECONDARY OUTCOMES:
Sleep quality | MOS Sleep Scale
Anxiety symptoms | 7 days, 6 weeks, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M McLean, MD MPH, Principal Investigator — UNC Chapel Hill School of Medicine
Locations (1):
- University of North Carolina Trauma Center, Chapel Hill, North Carolina, United States